CLINICAL TRIAL: NCT01341964
Title: Randomized Controlled Trial to Explore Interaction Between Aspirin and Clopidogrel in Stable Patients With Previous Myocardial Infarction or Coronary Artery Stent
Brief Title: Clopidogrel and Aspirin Interaction Study-2
Acronym: Interaction2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, John Eikelboom, Dr, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-090
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Drug Action Increased
Keywords: Clopidogrel; Aspirin; Interaction
MeSH Terms: interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher dose aspirin group (Experimental): Clopidogrel 600 mg plus aspirin 325mg
  Interventions: Drug: Clopidogrel; Drug: Aspirin
- Low dose aspirin group (Active Comparator): Clopidogrel 600mg plus aspirin 81mg
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 600mg (2 pills)
  Other Names: Plavix
Drug: Aspirin — 325mg (1 pill)
  Other Names: Novasen
  Arms: Higher dose aspirin group
Drug: Aspirin — 81mg (1 pill)
  Other Names: Entrophen
  Arms: Low dose aspirin group

SUMMARY:
Clopidogrel and aspirin are commonly used in combination to prevent heart attacks and to prevent blockage of stents. Both clopidogrel and aspirin work by preventing platelets (sticky cells that circulate in the blood) from forming blood clots in the arteries supplying oxygen to the heart and in stents. The investigators hypothesize that aspirin 325mg compared with aspirin 81 mg will increase blood levels of the active metabolite of clopidogrel in patients with a history of coronary artery disease who receive a 600mg loading dose of clopidogrel.

DETAILED DESCRIPTION:
Eligible patients will be randomized to receive clopidogrel 600mg + aspirin 325mg (Group A) or clopidogrel 600mg + aspirin 81mg (Group B). Patients will be fasted for at least 8 hours prior to study drug administration. Blood samples will be collected at 1 hour after study drug administration for measurement of clopidogrel active metabolite levels and genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients >1 month post ACS (including ST elevated myocardial infarction, non-ST elevated myocardial infarction or unstable angina) or stent
* Receiving regular ASA (81mg/d) and clopidogrel (75mg/d) for at least 1 week
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Liver disease with ALT or bilirubin >2x upper limits of normal (ULN)*
* Renal impairment with creatinine clearance <30 ml/min*
* Deemed to be at high risk of bleeding (e.g., recent bleeding, platelet count<100x109/L or hemoglobin <100g/L)*
* Anticoagulant or NSAID therapy within the last 5 days
* Antiplatelet agent other than aspirin and clopidogrel within the last 10 days
* Uncontrolled hypertension (>=180/110mmHg)

  * within 3 months of planned randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liang, MD, Principal Investigator — Population Health Research Institute; John Eikelboom, MD, Study Director — Population Health Research Institute
Locations (1):
- Population Health Research Institute, Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Liang Y, Hirsh J, Weitz JI, Sloane D, Gao P, Pare G, Zhu J, Eikelboom JW. Active metabolite concentration of clopidogrel in patients taking different doses of aspirin: results of the interaction trial. J Thromb Haemost. 2015 Mar;13(3):347-52. doi: 10.1111/jth.12829. Epub 2015 Feb 4. PMID 25557828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Higher Dose Aspirin Group | Low Dose Aspirin Group
Started | 152 | 150
Completed | 152 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with CAD on DAPT
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Dose Aspirin Group | Low Dose Aspirin Group | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 59.3 (9.3) | 61.5 (10.4) | 60.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 49 | 86
  Male | 115 | 101 | 216

OUTCOME MEASURES:

1. Primary Outcome: Blood Concentration of the Active Metabolite of Clopidogrel
Description: Clopidogrel active metabolite concentration will be measured by liquid chromatography tandem mass spectrometry (LC/MS) methods.
Time Frame: 1 hour after loading dose of study medications
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Clopidogrel Concentration of Higher Dose Aspirin Group: Clopidogrel 600 mg plus aspirin 325mg
  Clopidogrel: 600mg (2 pills)
  Aspirin: 325mg (1 pill)
- Clopidogrel Concentration of Low Dose Aspirin Group: Clopidogrel 600mg plus aspirin 81mg
  Clopidogrel: 600mg (2 pills)
  Aspirin: 81mg (1 pill)
Arm/Group | Clopidogrel Concentration of Higher Dose Aspirin Group | Clopidogrel Concentration of Low Dose Aspirin Group
Number analyzed (Participants) | 147 | 143
ng/ml | 14.45 [6.58 to 24.20] | 13.80 [7.62 to 20.20]
Statistical Analysis 1: Comparison: Clopidogrel Concentration of Higher Dose Aspirin Group vs Clopidogrel Concentration of Low Dose Aspirin Group; Test type: Superiority; p = 0.66, t-test, 2 sided; not normally distributed, values were log-transformed; Median Difference (Final Values) = 0.05

ADVERSE EVENTS:
Arm/Group | Clopidogrel Concentration of Higher Dose Aspirin Group | Clopidogrel Concentration of Low Dose Aspirin Group
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150
Other Adverse Events (participants affected / at risk) | 0/152 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No